CLINICAL TRIAL: NCT03633305
Title: Stepped Care Treatment for Insomnia Delivered in Primary Care Clinics: A Pragmatic Clinical Trial
Brief Title: Optimization of Insomnia Treatment in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Charles M. Morin, Professor, Laval University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIHR0083000212
Record Dates: First submitted 2018-07-17; First posted 2018-08-16 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Insomnia Disorder
Keywords: Insomnia; Pragmatic Clinical Trial; Drug Therapy; Cognitive Behavior Therapy; Primary Care
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Hypnotics and Sedatives

STUDY DESIGN:
Intervention Model Description: The study involves two treatment phases of six to eight weeks. In the first phase, participants choose medication (treatment as usual), online cognitive behavior therapy, or online cognitive behavior therapy combined with medication. Participants enter a second treatment phase if they still experience insomnia after the first treatment. The treatment arms for the second phase are medication, in-person cognitive-behavior therapy, or no additional treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment as usual (Active Comparator): Hypnotics - Medication used 1 to 7 nights/week for 6 to 8 weeks
  Interventions: Drug: Hypnotics
- Online cognitive behavior therapy (Experimental): Online CBT- Internet self-help program for insomnia with 6 cores
  Interventions: Behavioral: Online CBT
- Treatment as usual + Online CBT (Experimental): Hypnotics - Medication used 1 to 7 nights/week for 6 to 8 weeks Online CBT- Internet self-help program for insomnia with 6 cores
  Interventions: Drug: Hypnotics; Behavioral: Online CBT
- Medication (Experimental): Hypnotics - Medication used 1 to 7 nights/week for 6 to 8 weeks (arms 1, 3, 4)
  Interventions: Drug: Hypnotics
- In-person cognitive behavior therapy (Experimental): Face-to-face CBT- Face-to-face therapy with 3 to 4 individual sessions in a period of 6 to 8 weeks.
  Interventions: Behavioral: Face-to-face CBT
- No additional treatment (No Intervention)

INTERVENTIONS:
Drug: Hypnotics — Medication used 1 to 7 nights/week for 6 to 8 weeks.
  Arms: Medication; Treatment as usual; Treatment as usual + Online CBT
Behavioral: Online CBT — Internet self-help program for insomnia with 6 cores.
  Arms: Online cognitive behavior therapy; Treatment as usual + Online CBT
Behavioral: Face-to-face CBT — Face-to-face therapy with 3 to 4 individual sessions in a period of 6 to 8 weeks.
  Arms: In-person cognitive behavior therapy

SUMMARY:
The primary objective of this pragmatic clinical trial is to evaluate the efficacy, feasibility, and adaptability of pharmacological and non-pharmacological treatments for insomnia disorder, delivered in primary care clinics. The second objective is to evaluate the efficacy of a sequential (stepped care) approach for persistent insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Meeting criteria for insomnia disorder
* Registered patient at one of the primary care clinics participating in the study
* Fluent in French
* Computer and internet access

Exclusion Criteria:

* Unstable or untreated psychiatric disorder
* Lifetime psychotic or bipolar disorder
* Current suicide risk
* Progressive or unstable medical disorder
* Untreated sleep disorder other than insomnia
* Use of medication altering sleep
* Irregular or atypical sleep-wake schedule
* Current or planned pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Remission of insomnia | Post-1 (after 6-week treatment phase 1)
  Insomnia Severity Index score (average of two consecutive weeks < 8, with none > 10)
Remission of insomnia | Post-2 (after 6-week treatment phase 2)
  Insomnia Severity Index score (average of two consecutive weeks < 8, with none > 10)

SECONDARY OUTCOMES:
Total sleep time from sleep diary | Post-1 (after 6-week treatment phase 1)
  Mean total sleep time per night in minutes from sleep diary
Total sleep time from sleep diary | Post-2 (after 6-week treatment phase 2)
  Mean total sleep time per night in minutes from sleep diary
Total wake time from sleep diary | Post-1 (after 6-week treatment phase 1)
  Mean total wake time (combining sleep onset latency, wake after sleep onset, and duration of early morning awakening) in minutes from sleep diary
Total wake time from sleep diary | Post-2 (after 6-week treatment phase 2)
  Mean total wake time (combining sleep onset latency, wake after sleep onset, and duration of early morning awakening) in minutes from sleep diary
Sleep efficiency from sleep diary | Post-1 (after 6-week treatment phase 1)
  Mean sleep efficiency in percentage (total sleep time divided by time spent in bed, multiplied by 100) from sleep diary
Sleep efficiency from sleep diary | Post-2 (after 6-week treatment phase 2)
  Mean sleep efficiency in percentage (total sleep time divided by time spent in bed, multiplied by 100) from sleep diary
Total sleep time from actigraphy | Post-1 (after 6-week treatment phase 1)
  Mean total sleep time per night in minutes from actigraphy
Total sleep time from actigraphy | Post-2 (after 6-week treatment phase 2)
  Mean total sleep time per night in minutes from actigraphy
Total wake time from actigraphy | Post-1 (after 6-week treatment phase 1)
  Mean total wake time (combining sleep onset latency, wake after sleep onset, and duration of early morning awakening) in minutes from actigraphy
Total wake time from actigraphy | Post-2 (after 6-week treatment phase 2)
  Mean total wake time (combining sleep onset latency, wake after sleep onset, and duration of early morning awakening) in minutes from actigraphy
Sleep efficiency from actigraphy | Post-1 (after 6-week treatment phase 1)
  Mean sleep efficiency in percentage (total sleep time divided by time spent in bed, multiplied by 100) from actigraphy
Sleep efficiency from actigraphy | Post-2 (after 6-week treatment phase 2)
  Mean sleep efficiency in percentage (total sleep time divided by time spent in bed, multiplied by 100) from actigraphy
Fatigue | Post-1 (after 6-week treatment phase 1)
  Flinders Fatigue Scale (7-item self-report scale measuring fatigue over the past two weeks; total score ranges from 0 to 31, higher scores indicating greater fatigue)
Fatigue | Post-2 (after 6-week treatment phase 2)
  Flinders Fatigue Scale (7-item self-report scale measuring fatigue over the past two weeks; total score ranges from 0 to 31, higher scores indicating greater fatigue)
Depression | Post-1 (after 6-week treatment phase 1)
  Patient Health Questionnaire (PHQ-9)
Depression | Post-2 (after 6-week treatment phase 2)
  Patient Health Questionnaire (PHQ-9)
Anxiety | Post-1 (after 6-week treatment phase 1)
  Generalized Anxiety Disorder 7-item (GAD-7)
Anxiety | Post-2 (after 6-week treatment phase 2)
  Generalized Anxiety Disorder 7-item (GAD-7)
Disability | Post-1 (after 6-week treatment phase 1)
  Work and Social Adjustment Scale (5-item scale scale assessing functional impact of insomnia; total score ranging from 0 to 40, higher scores indicating greater disability)
Disability | Post-2 (after 6-week treatment phase 2)
  Work and Social Adjustment Scale (5-item scale scale assessing functional impact of insomnia; total score ranging from 0 to 40, higher scores indicating greater disability)
Medication use | Post-1 (after 6-week treatment phase 1)
  Frequency of use (number of nights/week)
Medication use | Post-2 (after 6-week treatment phase 2)
  Frequency of use (number of nights/week)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Morin, PhD, Principal Investigator — Université Laval Centre d'étude des troubles du sommeil
Locations (1):
- Laval University, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheung JMY, Ritterband LM, Chen SJ, Ivers H, Morin CM. Stepped-Care Management of Insomnia: Treatment Choices Guided by a Patient Decision Aid in a Pragmatic Nonrandomized Clinical Trial Setting. J Sleep Res. 2025 Jun 26:e70127. doi: 10.1111/jsr.70127. Online ahead of print. PMID 40570832
- [Derived] Morin CM, Chen SJ, Lemieux K, Ivers H, Cheung JMY, Lamy M, Ritterband L. Stepped care for insomnia in primary care using digital and face-to-face cognitive behavioral therapies: A pragmatic nonrandomized clinical trial. Sleep Med. 2025 Aug;132:106551. doi: 10.1016/j.sleep.2025.106551. Epub 2025 May 3. PMID 40373353